CLINICAL TRIAL: NCT02978131
Title: Evaluation of the Sensitivity of Histopathological Techniques and Molecular Biology (PCR) on Tissues Fixed in Paraformaldehyde and Included in Paraffin for the Diagnosis of Tuberculosis in Current Practice
Brief Title: Histopathological Techniques and PCR on Tissues Included in Paraffin for the Diagnosis of Tuberculosis
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-032
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Tuberculosis; Diagnostic Techniques and Procedures; Sensitivity and Specificity; Polymerase Chain Reaction; Immunohistochemistry; Histochemistry
Keywords: TUBERCULOSIS; Sensitivity and Specificity; Polymerase Chain Reaction; Immunohistochemistry; Histochemistry; Paraformaldehyde and paraffin embedded tissues
MeSH Terms: conditions — Tuberculosis; Hypersensitivity | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pulmonary and extrapulmonary, paraformaldehyde fixed and paraffin embedded tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a clinical diagnosis of TB: Patients with a clinical diagnosis of TB. Retrospective study on biopsy samples
  Interventions: Other: Histopathological study; Other: Molecular study (Polymerase chain reaction)

INTERVENTIONS:
Other: Histopathological study
Other: Molecular study (Polymerase chain reaction)

SUMMARY:
Tuberculosis (TB) remains a major public health problem nowadays. About 30% of the world population is infected with Mycobacterium tuberculosis. There is an increase in the number of cases of classic tuberculosis in developing countries, even if number of cases are declining in developed countries. However, in developed countries this decrease is counterbalanced by the emergence of multidrug resistant (MDR) strains of the bacteria.

There are also latent forms (1/3 of the world population) of the infection that can be reactivated in one case out of ten. Each year, about 2 million people die of tuberculosis and 9 million new cases are identified, including about 500,000 cases of MDR TB.

The spread of this disease as well as the increasing number of cases of MDR tuberculosis, reinforce the need for research and development of strategies of diagnosis and management of this affection.

Nowadays, the culture is the gold standard for the TB diagnosis but this technique needs at least three weeks to be performed. The objective of this study is to evaluate the sensitivity and specificity of histopathological and molecular techniques (PCR) on paraformaldehyde fixed and embedded in paraffin tissues for a faster diagnosis of tuberculosis in current practice, in order to administrate an efficient treatment as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Positive TB patients
* Patients who performed biopsy before inclusion

Exclusion Criteria:

* Anti-tuberculosis drugs administered before biopsy
* Patients who refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinical diagnosis of TB. Retrospective study on biopsy samples
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of positive TB cases with different techniques | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Colette Creusy, MD, Principal Investigator — GHICL

IPD SHARING:
Plan to Share IPD: No